CLINICAL TRIAL: NCT04548856
Title: Microsurgical Clipping and Endovascular Embolization Comparative Prospective Randomized Trial
Acronym: MONICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Boris Gegenava, Endovascolar surgery Chief, Moscow Regional Research and Clinical Institute (MONIKI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MONICA - Trial
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Ruptured Cerebral Aneurysm; Unruptured Cerebral Aneurysm
Keywords: Cerebral Aneurysm; Subarachnoid hemorrhage; Endovascular; Clipping; Embolization; Coiling
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: The stratified patients will be randomized into two groups (100 to the microsurgical clipping group and 100 to the endovascular embolization group). Each group will be divided into 2 subgroups of 50 people each: the first subgroup includes patients in the acute period of aneurysm rupture, the second subgroup includes patients with unruptured aneurysms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IA-Microsurgical clipping group (ruptured aneurysms) (Other): This subgroup includes patients who underwent microsurgical clipping of an acutely ruptured cerebral aneurysm
  Interventions: Procedure: Microsurgical clipping
- IB-Microsurgical clipping group (unruptured aneurysms) (Other): This subgroup includes patients who underwent microsurgical clipping of unruptured cerebral aneurysm
  Interventions: Procedure: Microsurgical clipping
- IIA-Endovascular embolization group (ruptured aneurysms) (Other): This subgroup includes patients who underwent endovascular embolization of an acutely ruptured cerebral aneurysm
  Interventions: Procedure: Endovascular embolization
- IIB-Endovascular embolization group (unruptured aneurysms) (Other): This subgroup includes patients who underwent endovascular embolization of unruptured cerebral aneurysm
  Interventions: Procedure: Endovascular embolization

INTERVENTIONS:
Procedure: Microsurgical clipping — Subjects randomized to surgical therapy will receive treatment from one neurosurgeon expert in surgery for ruptured aneurysms.
  Arms: IA-Microsurgical clipping group (ruptured aneurysms); IB-Microsurgical clipping group (unruptured aneurysms)
Procedure: Endovascular embolization — Subjects randomized to endovascular therapy will be treated by one endovascular expert in such treatment. Endovascular treatment will include all modern accepted surgical techniques.
  Arms: IIA-Endovascular embolization group (ruptured aneurysms); IIB-Endovascular embolization group (unruptured aneurysms)

SUMMARY:
Despite the active development of surgical methods of treatment (endovascular embolization and microsurgical clipping) of cerebral aneurysms, determining the indications and method of surgical treatment of cerebral aneurysms still causes debate in many cases. To a greater extent, this concerns the treatment of unruptured aneurysms. While there are a number of randomized trials of surgical treatment of ruptured cerebral aneurysms, there is currently no published randomized trial comparing surgical clipping and endovascular embolization of unruptured aneurysms. The purpose of this study is to compare the safety and efficacy of microsurgical clipping and endovascular embolization of cerebral aneurysms (both ruptured and unruptured) in a prospective, randomized fashion.

DETAILED DESCRIPTION:
The study is planned to include 200 patients. Before randomization, patients will be stratified according to the presence or absence of aneurysm rupture in the acute period. The stratified patients will be randomized into two groups (100 to the microsurgical clipping group and 100 to the endovascular embolization group). Each group will be divided into 2 subgroups of 50 people each: the first subgroup includes patients in the acute period of aneurysm rupture, the second subgroup includes patients with unruptured aneurysms. Patients will be followed postoperatively, outcome endpoints will be assessed at discharge, 6 and 12 months. At discharge and after 6 and 12 months, patients will be assessed clinically using a modified Rankin scale (mRS). Cerebral angiography will be performed intraoperatively (endovascular group), after surgery (microsurgical group) and 12 months after discharge (both groups). Thus, the outcome of surgical treatment, including periprocedural complications and mortality, will be assessed both clinically and angiographically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ruptured (acute SAH) or unruptured cerebral aneurysm who require surgical treatment (clipping and / or embolization)
* Both male and female
* Age from 18 to 80 years
* Informed consent to participate in the study signed by the patient. If the patient cannot give consent, informed consent is signed by closest relatives or based on the results of a medical concilium
* The patient (legal representative) agrees to a clinical assessment (examination and / or telephone visit) within 6 months and 12 months and to an angiographic control after 12 months
* Patient has not previously been randomized to this or other ongoing study
* Aneurysm has not previously been treated with endovascular embolization or microsurgical clipping

Exclusion Criteria:

* The target aneurysm has been treated (embolization or clipping) before
* Severe clinical condition of the patient (Glasgow coma scale <4, unstable hemodynamics)
* Lack of signed informed consent
* Severe medical or surgical comorbidity in which the patient's life expectancy is less than 2 years
* Pregnancy, breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2023-09-14 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) | 6 and 12 months after discharge
  Assessment of the clinical condition of patients will be carried out according to the modified Rankin scale (mRS). Primary Outcome Measure is modified Rankin Scale < or = to 2. mRS will be studied before surgery, after surgery, 6 and 12 months after discharge. Also the dynamics of changes in mRS compared with the baseline values will be analyzed. The null hypothesis is that no difference in outcome will be detected between the endovascular and surgical treatment arms. A statistically significant difference will then be considered evidence in favor of the alternative hypothesis, that one treatment is superior to the other.

SECONDARY OUTCOMES:
Death | 12 months
  Death associated with an underlying disease or its complication, or complication after surgery
Grading the occlusion of treated cerebral aneurysms | 12 months
  Assessed as total occlusion of the aneurysm or the presence of residual filling of the aneurysm
Aneurysm recanalization | 12 months
  Recanalization of the aneurysm after surgery will be assessed by cerebral angiography after 12 months
Reoperations | 12 months
  Additional operations on the target aneurysm after the initial intervention
Periprocedural complications | 12 months
  Any complications associated with surgical intervention: hematoma in the puncture area, dissection of arteries, postoperative intracranial hematoma, liquorrhea, postoperative meningitis, suppuration of postoperative stitches, neurological complications, etc.
Stroke | 12 months
  Ischemic or hemorrhagic stroke in the target artery